CLINICAL TRIAL: NCT01495897
Title: Adaptation Sensorimotrice, Cervelet et Mouvements Anormaux: Projet d'étude Oculomotrice
Brief Title: Abnormal Movements, Cerebellum and Sensorimotor : Oculomotor Study
Acronym: MOUVADOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C10-18; 2010-A00740-39 (Other: Afssaps)
Record Dates: First submitted 2011-05-18; First posted 2011-12-20 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2016-02

CONDITIONS: Healthy; Dystonia; Parkinson Disease
Keywords: Dystonia; Cerebellar; ocular movements; DYT 11; sensorimotor integration
MeSH Terms: conditions — Dystonia; Parkinson Disease | interventions — Eye-Tracking Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy (Other): Healthy volunteers
  Interventions: Device: Tracking eye movement
- Dystonia (Experimental): patients with Primary Dystonia
  Interventions: Device: Tracking eye movement
- Parkinson (Experimental): patients with Parkinson's disease
  Interventions: Device: Tracking eye movement
- Essential tremor (Experimental): patients with essential tremor with or without deep brain stimulation
  Interventions: Device: Tracking eye movement; Device: Tracking eye movement under deep brain stimulation

INTERVENTIONS:
Device: Tracking eye movement — Device: studying Saccadic eye movements with a video eye tracker: The subjects are seated in darkness facing a screen located 60 cm before their eyes, their chin on a chin strap and their forehead placed against a frontal support. Eye position is sampled at 500 Hz with a video-based monocular eye tracker (SMI, Germany). Each recording session start with a calibration test in which the subjects looked at nine consecutive targets covering the entire visual field, as used during the oculomotor paradigms: four experimental conditions: a visually guided saccade task, a pre-test, a backward adaptation task, and a post-test. The pre-test and post-test (40 trials each) are performed before and immediately after the backward adaptation task, in the same conditions, except that the target was extinguished when the velocity threshold (150°/s for 10 ms) is reached, instead of jumping to a new location.
Device: Tracking eye movement under deep brain stimulation — Device: studying Saccadic eye movements with a video eye tracker. If the patient has deep brain stimulation, recording will be made in the morning, before the usual morning start of the deep brain stimulation.
  Arms: Essential tremor

SUMMARY:
Dystonia is a movement disorder characterized by involuntary, sustained, often repetitive muscle contractions of opposite muscles that lead to abnormal twisting movements or odd postures. Essential tremor is a slowly progressive neurologic disorder characterized by the appearance of a tremor during the voluntary movement. The pathophysiology of dystonia or essential tremor is not fully elucidated. Dystonia and essential tremor are associated with dysfunction of the sensorimotor basal ganglia-cortical network and involvement of the cerebellum and cerebellar pathways has also been recently suggested.

The investigators propose to study 30 patients having a primary dystonia (15 DYT11 genetically documented), 15 patients having an essential tremor without deep brain stimulation and 15 patients having an essential tremor with deep brain stimulation.A group of 30 healthy volunteers will be recruited and tested according to the same modalities. They will be paired in sex and age. 30 patients having a Parkinson disease will be also tested.

Eye position will be sampled with a video-based monocular eye tracker (SMI, Germany) before and immediately after an adaptation task. Saccade adaptation is evaluated as the percentage change in the mean saccade amplitude between pre-test and post-test.

Expected results:

* no or fewer alteration of the performance to the adaptation task in the Parkinson group than in the Essential Tremor group/ dystonia group.
* abnormal reactive saccade backward adaptation in the Dystonia group and Essential Tremor group, providing further neurophysiological evidence of cerebellar dysfunction.

DETAILED DESCRIPTION:
Dystonia is a movement disorder characterized by involuntary, sustained, often repetitive muscle contractions of opposite muscles that lead to abnormal twisting movements or odd postures. Essential tremor is a slowly progressive neurologic disorder characterized by the appearance of a tremor during the voluntary movement. High frequency stimulation of the ventral intermedius nucleus (Vim) of the thalamus, relay for the cerebellar output, is successfully used for the treatment of severe essential tremor. It occasionally induces adverse event such as balance disorders or cerebellar symptoms. The pathophysiology of dystonia or essential tremor is not fully elucidated. Dystonia and essential tremor are associated with dysfunction of the sensorimotor basal ganglia-cortical network and involvement of the cerebellum and cerebellar pathways has also been recently suggested. It seems that dystonia and essential tremor could be the result of basal ganglia or cerebellar dysfunction, or from dysfunction of structures controlled at the same time by the cerebellum and the basal ganglia.

methodology: We propose to study 30 patients having a primary dystonia (15 DYT11 genetically documented), 15 patients having an essential tremor without deep brain stimulation and 15 patients having an essential tremor with deep brain stimulation.

A group of 30 healthy volunteers will be recruited and tested according to the same modalities. They will be paired in sex and age. 30 patients having a Parkinson disease will be also tested.

The subjects will be seated in darkness facing a screen located 60 cm before their eyes, their chin on a chin strap and their forehead placed against a frontal support. Eye position is sampled at 500 Hz with a video-based monocular eye tracker (SMI, Germany). Each recording session start with a calibration test in which the subjects looked at nine consecutive targets covering the entire visual field, as used during the oculomotor paradigms: four experimental conditions: a visually guided saccade task, a pre-test, a backward adaptation task, and a post-test. The pre-test and post-test (40 trials each) are performed before and immediately after the backward adaptation task, in the same conditions, except that the target was extinguished when the velocity threshold (150°/s for 10 ms) is reached, instead of jumping to a new location. This avoided any post-saccadic visual feedback that would counteract the adaptive mechanism. Saccade adaptation is evaluated as the percentage change in the mean saccade amplitude between the pre-test and post-test.

Expected results:

* no or fewer alteration of the performance to the adaptation task in the Parkinson group than in the Essential Tremor group/ dystonia group.
* abnormal reactive saccade backward adaptation in the Dystonia group and Essential Tremor group, providing further neurophysiological evidence of cerebellar dysfunction.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years
* -normal cognitive functions (>24y)
* Normal clinical examination of ocular mobility, visualization of the target
* No drug potentially able to modify and to influence the data: anti-depressants, neuroleptics, anti-emetics, amphetamines, anti myoclonic/dystonic drugs, alcohol, dopaminergic drug, antiepileptic.
* Dystonia or essential tremor or Parkinson: diagnostic made by a neurologist
* For DYT11: mutation in SGCE gene.
* For dystonia: No secondary dystonia
* For Parkinson : UPDRS<28
* No other neurological disorder

For the patient having deep brain stimulation:

* Duration of stimulation> 6 months
* Cerebral imagery post operation made
* Stimulation parameter stable since 3 months at least.
* Usual stop of the stimulation during the night

Exclusion criteria:

* Uncontrollable medical problems not related to M-D
* Current active psychiatric disorder
* Intake during the last 3 days of drugs potentially able to modify and to influence the data: anti-depressants, neuroleptics, anti-emetics, amphetamines, anti myoclonic/dystonic drugs, alcohol, dopaminergic drug
* Subjects legally protected.
* Subjects who are not enrolled at social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Saccadic adaptation | between the pre-test and post-test, maximum 4 hours
  Saccadic adaptation, evaluated as the percentage of changes in the mean saccade amplitude between the pre-test and post-test.
Characteristics of the saccade | measured during the analysis of the recorded session, maximum 4 hours
  latency, velocity, duration of the saccade

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Flamand-Roze, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- : Fédération des Maladies du Système Nerveux, Paris, France

REFERENCES:
- [Background] Hubsch C, Vidailhet M, Rivaud-Pechoux S, Pouget P, Brochard V, Degos B, Pelisson D, Golmard JL, Gaymard B, Roze E. Impaired saccadic adaptation in DYT11 dystonia. J Neurol Neurosurg Psychiatry. 2011 Oct;82(10):1103-6. doi: 10.1136/jnnp.2010.232793. Epub 2011 Mar 8. PMID 21386109